CLINICAL TRIAL: NCT00272818
Title: Non-Invasive Markers in the Diagnosis and Interval Assessment of Children and Adults With Known or Suspected Allergic Disease
Brief Title: Study to Identify Non-Invasive Markers of Gastrointestinal Allergy
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: TechLab, Incorporate (Other)
Responsible Party: Principal Investigator, Web, Assistant Professor of Pediatrics, Boston Children's Hospital
Other Study IDs: 04-07-042
Record Dates: First submitted 2006-01-04; First posted 2006-01-09 (Estimated); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Esophagitis; Colitis
Keywords: Colitis; Esophagitis; CD23
MeSH Terms: conditions — Esophagitis; Colitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The incidence of gastrointestinal allergy is on the rise and can be manifest in a number of different clinical presentations. The goal of this study is to evaluate the measurement of CD23, a protein that can be identified stool, urine, and blood, as a non-invasive marker for use in the diagnosis and interval assessment of patients with known or suspected gastrointerstianl allergy.

Eosinophilic esophagitis (EE) is a disorder typically found in school-age and adolescent children, and is more prevalent in male patients. Patients with EE typically present with symptoms of heartburn or difficulties swallowing. Blood and x-ray studies may be normal or display non-specific findings. The diagnosis of EE rests on a combination of clinical symptoms, and the results of endoscopic and histologic studies. There is currently no biochemical marker that can be used to monitor disease course in these patients.

Cow milk protein intolerance (CMPI) is an allergic process affecting the distal gastrointestinal tract in infants. As such, it often presents as diarrhea without or without the presence of gross rectal bleeding in infants ranging in age from birth to 6 months of age. Children display symptoms of abdominal disress including emesis, cramping, colic, or feeding difficulties. The diagnosis is based on an appropriate clinical history and supporting physical exam (typically normal). Treatment involves removal of the offending dietary antigens which include cow or soy milk protein Eosinophilic crypt abscesses, or collections of eosinophils within the intestine can also be seen.

CD23 is a protein that can be found on allergy-type white blood cells (eosinophils), as well as on the cells that line the gastrointestinal tract. Previous studies have reported increased levels of CD23 in infants with cow's milk allergy. CD23 is also elevated in infants and children with allergic disease. Levels of CD23 appears to fall in conjunction with therapy.

DETAILED DESCRIPTION:
The incidence of gastrointestinal allergy is on the rise and can be manifest in a number of different clinical presentations. The goal of this study is to evaluate the measurement of CD23, a protein that can be identified stool, urine, and blood, as a non-invasive marker for use in the diagnosis and interval assessment of patients with known or suspected gastrointerstianl allergy.

Eosinophilic esophagitis (EE) is a disorder typically found in school-age and adolescent children, and is more prevalent in male patients. Patients with EE typically present with symptoms of heartburn or difficulties swallowing. Blood and x-ray studies may be normal or display non-specific findings. The diagnosis of EE rests on a combination of clinical symptoms, and the results of endoscopic and histologic studies. The endoscopic appearance of esophageal mucosa in these patients is often pale and displays a poor vascular pattern. The mucosa can be thickened in appearance. Esophagitis in patients with acid/peptic disease is typically more pronounced at the bottom of the esophagus, in the region of the gastroesophageal junction. In contrast, the mucosal disease observed in patients with EE is often more pronouced in the proximal esophagus. Treatment may include topial steroids (delivered systemically or via metered-dose inhaler) and formal allergy evaluation to detect potential dietary triggers. Anti-allergic therapies, including monteleukostat, benedryl, antihistimines, and cromolyn sodium have also been proposed as treatments for EE. Treatment efficacy is determined by a combination of clinical report and serial endoscopic study. There is currently no biochemical marker that can be used to monitor disease course in these patients.

Cow milk protein intolerance (CMPI) is an allergic process affecting the distal gastrointestinal tract in infants. As such, it often presents as diarrhea without or without the presence of gross rectal bleeding in infants ranging in age from birth to 6 months of age. Children display symptoms of abdominal disress including cramping, colic, or feeding difficulties. Emesis after feeds may also be present. Affected children display loose and more frequent bowel movements. Stools in these patients may contain mucus as well as microscopic or visible blood. In most patients, the diagnosis is based on an appropriate clinical history and supporting physical exam (typically normal). Treatment involves removal of the offending dietary antigens which include cow or soy milk protein. A small percentage of patients (< 5%) require formal endoscopic study. The mucosa in these patients appears erythematous, friable, and can display a patchy distribution of inflammation. Histologic exam reveals varying degrees of eosinophic infiltration of the intestinal tissue. Eosinophilic crypt abscesses, or collections of eosinophils within the intestine can also be seen. Patients responding to therapy will display normalization of stool frequency, decreased symptoms of abdominal discomfort, and an absence of gross or microscopic intestinal bleeding.

CD23 is a protein that can be found on allergy-type white blood cells (eosinophils), as well as on the cells that line the gastrointestinal tract. Previous studies have reported increased levels of CD23 in infants with cow's milk allergy. CD23 is also elevated in infants and children with allergic disease, when compared to to children without apparent atopic disease. Moreover, the level of CD23 appears to fall in conjunction with therapy.

The development of non-invasive markers of intestinal allergy would facilitate diagnosis as well as provide clinicians with a tool to assess patients compliance and response to therapy. The relationship between levels of serum, urinary, and fecal CD23 levels has not been previously studied in patients with known or suspected intestinal allergy.

Subjects in this study will be asked to provide a blood, urine, and stool sample when they present with symptoms or either cow milk protein intolerance or eosinophilic esophagitis. Blood will only be obtained if clinical samples are requested, and no extra blood drawing will be required for participation in this study. Similar blood, urine, and stool specimens will be obtained after the patient has been placed on anti-atopic therapy and is experiencing clinical remission.

ELIGIBILITY:
Inclusion Criteria:

Known or suspected cow milk protein intolerance Known or suspected eosinophilic esophagitis

Exclusion Criteria:

None

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients with known or suspected GI allergy.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2004-09; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul A. Rufo, MD, MMSc, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital, Boston, Massachusetts, United States